CLINICAL TRIAL: NCT06146192
Title: Withdrawal of Colchicine in Behçet Syndrome Patients With Skin and Mucosa Involvement
Brief Title: Withdrawal of Colchicine in Behçet Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulen Hatemi, Professor, Istanbul University - Cerrahpasa
Other Study IDs: 431693
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Behçet's Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — Colchicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Colchicine
  Interventions: Drug: Colchicine
- No colchicine

INTERVENTIONS:
Drug: Colchicine — colchicine 1-2 mg/day
  Groups: Colchicine

SUMMARY:
Behçet's syndrome is a multisystem variable vessel vasculitis. Clinical features include mucocutaneous manifestions such as oral ulcers, genital ulcers, papulopustular lesions and nodular lesions, musculoskeletal manifestations, uveitis, venous thrombosis, arterial aneurysms and thrombosis, central nervous system involvement and gastrointestinal involvement. Management of Behçet's syndrome depends on the type of organ involvement, disease severity, and prognostic factors. The main objective in patients with major organ involvement is to rapidly suppress the inflammation and prevent relapses in order to prevent organ damage. On the other hand, mucocutaneous and musculoskeletal manifestations do not cause damage and in patients with only mucocutaneous and joint involvement, the aim is to improve the quality of life.

Colchicine is usually the first-line systemic treatment in patients with only mucocutaneous and joint involvement. Conflicting results were reported on the efficacy of colchicine on different mucocutaneous manifestations in randomized placebo-controlled trials. The relapsing and remitting nature of these manifestations in Behçet's syndrome may cause challenges in disease assessment during clinical trials. Another approach to evaluate the effectiveness of a medication is to evaluate whether the lesions recur or increase after discontinuation of the drug. The aim of this study is to assess mucocutaneous disease activity among Behçet's syndrome patients after discontinuation of colchicine treatment and compare it to patients who continue to use colchicine.

ELIGIBILITY:
Inclusion Criteria:

Fulfilling International Study Group criteria. Being between the ages of 18 and 65 years. Having mucocutaneous involvement. Using colchicine at a stable dose (1-2 mg/day) for at least 3 months. Showing no adverse events related to colchicine use. Providing informed consent to participate in the study. -

Exclusion Criteria:

Patients with active uveitis. Patients with active venous involvement. Patients with active arterial involvement. Patients with active nervous system involvement. Patients with active gastrointestinal involvement.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Behçet's syndrome patients with mucocutaneous involvement who have been using colchicine at a stable dose (1-2 mg/day) during the last 3 months and who do not have any active organ involvement (ie uveitis, venous thrombosis, arterial aneurysms or thrombosis, nervous system involvement, and gastrointestinal involvement).
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of oral ulcers | 4 weeks

SECONDARY OUTCOMES:
Number of genital ulcers | 4 weeks
Number of nodular lesions | 4 weeks
Pain of oral ulcers | 4 weeks
Pain of genital ulcers | 4 weeks
Pain of nodular lesions | 4 weeks
Number of papulopustular lesions | 4 weeks
Tender joint count | 4 weeks
Swollen joint count | 4 weeks
Overall disease activity | 4 weeks
  Overall disease activity will be assessed using Behçet's disease current activity form and Behçet's syndrome activity scale
Health related quality of life | 4 weeks
  Health related quality of life will be assessed using short form 36 V2 and Behçet's disease quality of life scale
New organ involvement | 4 weeks

IPD SHARING:
Plan to Share IPD: Yes